CLINICAL TRIAL: NCT04278027
Title: Epigenetic Regulation of Brain-Derived Neurotrophic Factor (BDNF) Gene Expression According to Response to Cognitive Remediation in Schizophrenia
Brief Title: Cognitive Remediation Therapy in Schizophrenia: Effects on Epigenetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Rafael Penades, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24618; PI17/00872 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
Keywords: Cognitive Remediation; Epigenetics; BDNF
MeSH Terms: conditions — Schizophrenia | interventions — Gene Regulatory Networks

STUDY DESIGN:
Intervention Model Description: Study Procedure. 60 patients with schizophrenia disorder (according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) classification, determined by The Structured Clinical Interview for DSM-5 (SCID-5) interview will be recruited and randomly allocated in one of the two groups: CRT or treatment as usual control group. All participants will undergo neurocognitive testing over a 2-week period, followed by a blood draw. After random allocation, 40 participants will follow a computerized cognitive remediation program and 20 will be followed a similar period of time without any cognitive intervention. Subjects will have another blood sample drawn after completion of the cognitive therapy or the TAU. All subjects should remain on stable doses of medications while in the study (no dose change > 10%). Finally, subjects will be reassessed on PANSS and cognitive measures and social functioning by personnel blind to group assignment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation Therapy (Experimental): Cognitive Remediation Therapy. CRT will be based on CIRCuiTS, a computerized program.
  Interventions: Behavioral: Cognitive Remediation Therapy
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — "CIRCuiTS is a web-based computerised CR therapy, delivered by a therapist but supplemented with independent sessions to facilitate massed practice. It targets metacognition, particularly strategy use, in addition to providing massed practice of basic cognitive functions. The therapist facilitates motivation, metacognitive and strategy development and generalisation of learning by encouraging the participant to learn about and regulate their cognitive performance and to transfer this learning to meet real-world goals. Therapists provide additional scaffolding for CR tasks to ensure consistent successful performance. Independent sessions involve carrying out cognitive tasks allocated by the therapist to ensure scaffolded learning" (Reeder et al.2017)
  Other Names: CIRCuiTS
  Arms: Cognitive Remediation Therapy

SUMMARY:
This study is a randomised and controlled trial that aims to investigate whether Cognitive Remediation Therapy (CRT) can modulate epigenetic mechanisms by changing methylation levels of BDNF gene in patients with Schizophrenia.

DETAILED DESCRIPTION:
OBJECTIVES: To investigate whether Cognitive Remediation Therapy (CRT) can modulate epigenetic mechanisms by changing methylation levels of BDNF gene. It also aims to test whether BDNF valine-66-methionine (Val66Met) polymorphism influences CRT treatment outcome among people with schizophrenia.

SAMPLE AND METHODS: A randomized and controlled study will be carried out with two groups: patients receiving CRT and patients in control condition without any cognitive intervention and receiving Treatment as Usual (TAU). Methylation levels of BDNF gene at different sites will be contrasted before and after treatment. Additionally, neurocognition profile, level of symptoms and psychosocial functioning will also be tested. CRT outcomes will be investigated in a mixed model for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-5 and confirmed by the semi-structured interview (SCID) for the axis 1.
* Presence of cognitive impairment confirmed by the neuropsychological battery
* Stable symptomatology at least during the last six months and the estimation of not modifying pharmacological antipsychotic treatment .

Exclusion Criteria:

* Presence of organic-cerebral affectation due to neurological or traumatic conditions
* Antipsychotic dose change >10%
* Abuse of psychotropic substances
* Presence of other psychiatric symptomatology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in methylation at Cytosine-phosphate-Guanine (CpG) exon | Baseline and after 4 months
  Mean methylation percentage in CpG island BDNF CpG exon I: located at chr11:27743473-27744564 in the BDNF
Change in methylation at CpG exon IV | Baseline and after 4 months
  Mean methylation percentage of CpG region BDNF CpG exon IV: located at chr11:27723060-27723294 in exon IV, upstream of the start codon in exon VII

SECONDARY OUTCOMES:
Change in cognition | Baseline and after 4 months
  Total score in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Change in Symptoms | Baseline and after 4 months
  Total score in Positive and Negative Syndromes Scale (PANSS)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Penadés, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Penades R, Almodovar-Paya C, Garcia-Rizo C, Ruiz V, Catalan R, Valero S, Wykes T, Fatjo-Vilas M, Arias B. Changes in BDNF methylation patterns after cognitive remediation therapy in schizophrenia: A randomized and controlled trial. J Psychiatr Res. 2024 May;173:166-174. doi: 10.1016/j.jpsychires.2024.03.014. Epub 2024 Mar 23. PMID 38537483